CLINICAL TRIAL: NCT03415490
Title: Folded and Classic Techniques of Self-adherent Wrap for Eyes After Orbital Tumour Extirpation
Brief Title: Self-adherent Wrap Techniques for Orbital Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201801
Record Dates: First submitted 2018-01-18; First posted 2018-01-30 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Surgery; Eye Diseases
Keywords: general anesthesia; self-adherent wrap; pressure
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic technique of self-adherent wrap (Active Comparator): 1. over 16 years old
  2. free of any symptoms in the eyes
  3. classic technique of self-adherent wrap after surgery
  Interventions: Other: Classic technique of self-adherent wrap
- Folded technique of self-adherent wrap (Experimental): 1. over 16 years old
  2. free of any symptoms in the eyes
  3. folded technique of self-adherent wrap after surgery
  Interventions: Other: Folded technique of self-adherent wrap

INTERVENTIONS:
Other: Folded technique of self-adherent wrap — Wrapping a piece of self-adherent wrap around the patient's head starting with the opened end on the forehead above the affected eye.The bandage is then firmly but not tightly wrapped around the head twice. Then, after the second circuit, the bandage is brought on the cheek and up over the eye to the forehead, where it was passed between the eyebrows but not wrapped around the head. Instead, the bandage is folded and then first passed back on the cheek of the affected side then back to the forehead a total of four times. Finally, the bandage is wrapped completely around the head once
  Arms: Folded technique of self-adherent wrap
Other: Classic technique of self-adherent wrap — Wrapping a piece of self-adherent wrap around the patient's head starting with the opened end on the forehead above the affected eye.The bandage is then firmly but not tightly wrapped around the head twice. After the second circuit, the bandage was brought below the ear, up over the eye and around the head of the non-affected side and then wrapped around the head in the same manner four times. The bandage is then brought around the head once.
  Arms: Classic technique of self-adherent wrap

SUMMARY:
The purpose of this study is to evaluate the interface pressure measurements of applying self-adherent wraps on eyes after orbital tumour extirpation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the interface pressure measurements of the folded and classic techniques of applying self-adherent wraps on eyes after orbital tumour extirpation.

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old
* diagnosed as orbital disease or ocular tumor
* surgery under general anesthesia

Exclusion Criteria:

* any uncontrolled clinical problems

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-21 (Actual)

PRIMARY OUTCOMES:
the pressure on the affected eye | 10 minutes after bandage application in awake individuals
  the pressure on the affected eye using the two methods

SECONDARY OUTCOMES:
the pressure outside the affected eye | 10 minutes after bandage application in awake individuals
  the pressure outside the affected eye using the two methods
discomfort scores | 1 minute after recording the pressures
  Discomfort levels were measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no discomfort and 10 represents the worst discomfort; this scale has been confirmed to be sensitive and reliable. Discomfort was defined as "sensation other than pain" and included nausea, vomiting, headache, and dizziness. Clinically significant postoperative discomfort was considered serious discomfort (NRS score ≥5) any time postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye Ye, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No